CLINICAL TRIAL: NCT06094894
Title: Changes in Gut Microbiota and Postprandial GLP-1 Concentration Due to Sucralose Consumption
Brief Title: Effects of Sucralose in Gut Intestinal Microbiota and Postprandial GLP-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Principal Investigator, Paloma Almeda-Valdés, MD, PhD, Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 2635.2
Record Dates: First submitted 2023-10-17; First posted 2023-10-23 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: GLP-1; Gut Microbiota; Insulin Resistance
Keywords: incretins; gut microbiota; sucralose; insulin resistance
MeSH Terms: conditions — Insulin Resistance | interventions — trichlorosucrose

STUDY DESIGN:
Intervention Model Description: Triple blind parallel placebo-controlled randomized clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The use of identical capsules will allow the blinding, the capsules will be deposited in bottles numbered sequentially according to the enrollment process and neither the participants nor the researchers will know the content of the capsules, or the group assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sucralose (Experimental): The intervention will consist of capsules filled with pure sucralose. Each capsule will contain 90 mg of sucralose. Participants will be asked to consume one capsule in each meal (three per day) to achieve an ingestion of 270 mg of sucralose, this quantity corresponds approximately to the 30% of the acceptable daily intake (ADI) of sucralose for a lean person. This was calculated based on the ADI established by the joint FAO/WHO expert committee on food additives (JECFA) of 15 mg per kg of body weight per day of sucralose.
  Interventions: Other: sucralose
- Placebo (Placebo Comparator): The intervention will consist of capsules filled with placebo (cornstarch). Each capsule will contain 90 mg of cornstarch. Participants will be asked to consume one capsule in each meal (three per day) in order to achieve an ingestion of 270 mg of placebo, this quantity is in order to match the sucralose consumed in the intervention group.
  Interventions: Other: placebo

INTERVENTIONS:
Other: sucralose — Food additive used to replace sugar providing a sweet taste without calories.
  Other Names: non-nutritive sweetener
  Arms: Sucralose
Other: placebo — Cornstarch without significant physiological effects
  Arms: Placebo

SUMMARY:
Recently, it has been proposed that the consumption of non-nutritive sweeteners, including sucralose, it's not harmless and is related with metabolic effects. Some studies have reported that sucralose produces alterations in glucose homeostasis. In vitro studies indicate that sucralose can interact with sweet taste receptors (T1R2 and T1R3) in the intestine, thus increasing the expression of glucose transporters including the sodium-glucose cotransporter type 1 (SGLT1) and the glucose transporter 2 (GLUT2), increasing glucose absorption. This interaction with intestinal sweet taste receptors also generates an increase in the secretion of the incretins glucagon-like peptide type 1 (GLP-1) and the glucose-dependent insulinotropic polypeptide (GIP), which might enhance the postprandial insulin release. However, these results are preliminary and it's desirable to confirm if sucralose consumption is associated with glucose metabolism modifications using an appropriate methodological design and with gold standard methods. The aim of this triple-blind, placebo-controlled, parallel, randomized clinical trial is to confirm the changes in insulin sensitivity associated with sucralose consumption in humans, to identify whether these changes are in the liver or skeletal muscle and to investigate the pathophysiological mechanisms generating these changes. Specifically, we will investigate if sucralose generates a dysbiosis in the gut microbiota that could be related to insulin resistance by increasing concentrations of lipopolysaccharide, a toxin found in Gram-negative bacteria that triggers a low-grade inflammation known as metabolic endotoxemia. In addition, the changes in postprandial concentrations of GLP-1, glucose, insulin, and C-peptide due to the combination of sucralose with a mixed meal will be investigated. The results of this study will determine if sucralose consumption, frequently used as a non-nutritive sweetener, is associated to significant changes in glucose homeostasis in humans.

DETAILED DESCRIPTION:
Study design:

This is a triple-blind, parallel, placebo-controlled, randomized clinical trial.

Sample size:

The sample size was calculated to observe a difference of 20% in the Matsuda index between groups.

The calculation was done considering a probability of type I error (α) of 5%, with a power of 80% and adding an extra-20% for potential losses at follow-up.

The estimated sample size for the study is 40 subjects, 20 per group.

Randomization:

The participants will be randomly assigned to one of the two groups (sucralose or placebo) using the website Randomization.com (http://www.randomization.com) with a balanced block design of 5 blocks with 8 subjects each. The random allocation sequence will be done by an external researcher.

Intervention:

The intervention will consist of capsules filled with pure sucralose or placebo (cornstarch) accordingly to the group assignment. Each capsule will contain 90 mg of sucralose or placebo. Participants will be asked to consume one capsule in each meal (three per day) in order to achieve an ingestion of 270 mg of sucralose or placebo, this quantity corresponds approximately to the 30% of the acceptable daily intake (ADI) of sucralose for a lean person. This was calculated based on the ADI established by the joint Food and Agriculture Organization of the United Nations (FAO)/World Health Organization (WHO) expert committee on food additives (JECFA) of 15 mg per kg of body weight per day of sucralose.

The use of identical capsules will allow the blinding, the capsules will be deposited in bottles numbered sequentially according to the enrollment process and neither the participants nor the researches will know the content of the capsules or the group assigned.

Visit 1

An oral glucose tolerance test (OGTT) will be performed to confirm that participants do not have diabetes or prediabetes. Fasting insulin, lipid profile and glycated hemoglobin will be measured. Also, anthropometry (weight, height, waist, and hip circumference), blood pressure and heart rate will be documented. Body composition will be evaluated with dual X-ray absorptiometry (DXA) already available in the Research Unit and bioelectrical impedance. Physical activity will be registered with the questionnaire from the University of Laval that measure energy expenditure in Kcal per day. A format for three-day food intake record will be given to be prospectively registered by participants.

Visit 2

The three-day food record will be requested and reviewed to evaluate food consumption habits. A mixed meal tolerance test will be performed over two hours. The meal will consist of 523 kcal (49% carbohydrates, 17% protein, 34% lipids). Blood samples will be collected at 0, 30, 60, 90 and 120 minutes to measure glucose, insulin and glucagon-like peptide type 1 (GLP-1) concentrations. Also, lipopolysaccharide (LPS), C-reactive protein (CRP), interleukin 6 (IL-6), and tumor necrosis factor-alpha (TNF-α) concentrations will be measured at the basal time. Ten minutes before the test participants will consume a capsule containing either sucralose or placebo (120 mg).

Participants will proportionate the first stool sample to evaluate gut microbiota.

The researchers will proportionate the bottle with capsules that each participant will consume during the intervention period (30 ± 2 days) in this visit. Also, each participant will be asked to record on the adherence format if they consumed the capsule at breakfast, lunch, and dinner each day of the intervention period and to record any symptom related to capsules ingestion. Another format to record three-day food consumption again will be given.

Visit 3

Participants will proportionate the second stool sample to evaluate changes in gut microbiota. Also, the physical activity questionnaire will be applied again, and the second 3-day food record will be obtained to evaluate changes in physical activity and food habits, respectively. The second mixed meal tolerance test will be performed following the same procedures as visit 2. Participants will be asked to return the empty bottles to quantify adherence to the intervention. In addition, adherence and symptoms formats will be collected.

Visit 4

Participants will be asked to assist one month after visit 3 to make a final evaluation of fasting glucose, insulin, and lipid profile concentrations. The physical activity questionnaire will be applied again, and a third 3-day food record will be collected to evaluate changes in physical activity and food habits, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Normal BMI (18.5-24.9 kg/m2)
* Low habitual consumption of non-nutritive sweeteners (NNS
* Fasting plasma insulin concentration of <12 mU/L

Exclusion Criteria:

* Diabetes or altered glucose metabolism (abnormal fasting glucose, glucose intolerance or elevated glycated hemoglobin)
* Use of antibiotics in the last 3 months
* Use of probiotics through pharmaceutical products
* Liver or kidney disease
* Use of medications that could interfere with insulin sensitivity
* Severe intestinal diseases
* History of bariatric surgery
* Pregnancy or lactation

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
glucose | baseline and 30 days after the intervention
  To evaluate the changes in postprandial glucose concentrations during a mixed meal after sucralose consumption in comparison to placebo
insulin | baseline and 30 days after the intervention
  To evaluate the changes in postprandial insulin concentrations during a mixed meal after sucralose consumption in comparison to placebo
C-peptide | baseline and 30 days after the intervention
  To evaluate the changes in postprandial C-peptide concentrations during a mixed meal after sucralose consumption in comparison to placebo
GLP-1 | baseline and 30 days after the intervention
  To evaluate the changes in postprandial GLP-1 area under the curve during a mixed meal after sucralose consumption in comparison to placebo
gut microbiota | baseline and 30 days after the intervention
  To compare the change in the relative abundance of colony forming units of bacterial genus and species after sucralose consumption in comparison to placebo through messenger RNA sequencing
PYY | baseline and 30 days after the intervention
  To evaluate the changes in postprandial PYY area under the curve during a mixed meal after sucralose consumption in comparison to placebo
ghrelin | baseline and 30 days after the intervention
  To evaluate the changes in postprandial ghrelin area under the curve during a mixed meal after sucralose consumption in comparison to placebo

SECONDARY OUTCOMES:
lipopolysaccharide | baseline and 30 days after the intervention
  To determine the effects of sucralose consumption in lipopolysaccharide concentrations in comparison to placebo
C-reactive protein | baseline and 30 days after the intervention
  To determine the effects of sucralose consumption in C-reactive protein concentrations in comparison to placebo
IL-6 | baseline and 30 days after the intervention
  To determine the effects of sucralose consumption in IL-6 concentrations in comparison to placebo
tumor necrosis factor-alpha | baseline and 30 days after the intervention
  To determine the effects of sucralose consumption in tumor necrosis factor-alpha concentrations in comparison to placebo

OTHER OUTCOMES:
fecal short chain fatty acids | baseline and 30 days after the intervention
  To determine the effects of sucralose consumption in fecal short chain fatty acids concentrations in comparison to placebo
serum fatty acid profile | baseline and 30 days after the intervention
  To determine the effects of sucralose consumption in serum fatty acid profile concentrations in comparison to placebo
Curli protein fecal expression | baseline and 30 days after the intervention
  To determine the effects of sucralose consumption in Curli protein fecal expresion concentrations in comparison to placebo
plasma branched-chain aminoacids | baseline and 30 days after the intervention
  To determine the effects of sucralose consumption in plasma branched-chain aminoacids concentrations in comparison to placebo

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Nacional de Ciencias Médicas y Nutrición Salvador Zubirán, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pepino MY, Tiemann CD, Patterson BW, Wice BM, Klein S. Sucralose affects glycemic and hormonal responses to an oral glucose load. Diabetes Care. 2013 Sep;36(9):2530-5. doi: 10.2337/dc12-2221. Epub 2013 Apr 30. PMID 23633524
- [Background] Romo-Romo A, Aguilar-Salinas CA, Gomez-Diaz RA, Brito-Cordova GX, Gomez-Velasco DV, Lopez-Rocha MJ, Almeda-Valdes P. Non-Nutritive Sweeteners: Evidence on their Association with Metabolic Diseases and Potential Effects on Glucose Metabolism and Appetite. Rev Invest Clin. 2017 May-Jun;69(3):129-138. doi: 10.24875/ric.17002141. PMID 28613282
- [Background] Suez J, Korem T, Zeevi D, Zilberman-Schapira G, Thaiss CA, Maza O, Israeli D, Zmora N, Gilad S, Weinberger A, Kuperman Y, Harmelin A, Kolodkin-Gal I, Shapiro H, Halpern Z, Segal E, Elinav E. Artificial sweeteners induce glucose intolerance by altering the gut microbiota. Nature. 2014 Oct 9;514(7521):181-6. doi: 10.1038/nature13793. Epub 2014 Sep 17. PMID 25231862
- [Background] Romo-Romo A, Aguilar-Salinas CA, Brito-Cordova GX, Gomez-Diaz RA, Almeda-Valdes P. Sucralose decreases insulin sensitivity in healthy subjects: a randomized controlled trial. Am J Clin Nutr. 2018 Sep 1;108(3):485-491. doi: 10.1093/ajcn/nqy152. PMID 30535090
- [Background] Lertrit A, Srimachai S, Saetung S, Chanprasertyothin S, Chailurkit LO, Areevut C, Katekao P, Ongphiphadhanakul B, Sriphrapradang C. Effects of sucralose on insulin and glucagon-like peptide-1 secretion in healthy subjects: a randomized, double-blind, placebo-controlled trial. Nutrition. 2018 Nov;55-56:125-130. doi: 10.1016/j.nut.2018.04.001. Epub 2018 Apr 21. PMID 30005329
- [Background] Dalenberg JR, Patel BP, Denis R, Veldhuizen MG, Nakamura Y, Vinke PC, Luquet S, Small DM. Short-Term Consumption of Sucralose with, but Not without, Carbohydrate Impairs Neural and Metabolic Sensitivity to Sugar in Humans. Cell Metab. 2020 Mar 3;31(3):493-502.e7. doi: 10.1016/j.cmet.2020.01.014. PMID 32130881
- [Background] Suez J, Cohen Y, Valdes-Mas R, Mor U, Dori-Bachash M, Federici S, Zmora N, Leshem A, Heinemann M, Linevsky R, Zur M, Ben-Zeev Brik R, Bukimer A, Eliyahu-Miller S, Metz A, Fischbein R, Sharov O, Malitsky S, Itkin M, Stettner N, Harmelin A, Shapiro H, Stein-Thoeringer CK, Segal E, Elinav E. Personalized microbiome-driven effects of non-nutritive sweeteners on human glucose tolerance. Cell. 2022 Sep 1;185(18):3307-3328.e19. doi: 10.1016/j.cell.2022.07.016. Epub 2022 Aug 19. PMID 35987213
- [Background] Bueno-Hernandez N, Esquivel-Velazquez M, Alcantara-Suarez R, Gomez-Arauz AY, Espinosa-Flores AJ, de Leon-Barrera KL, Mendoza-Martinez VM, Sanchez Medina GA, Leon-Hernandez M, Ruiz-Barranco A, Escobedo G, Melendez G. Chronic sucralose consumption induces elevation of serum insulin in young healthy adults: a randomized, double blind, controlled trial. Nutr J. 2020 Apr 13;19(1):32. doi: 10.1186/s12937-020-00549-5. PMID 32284053
- [Derived] Romo-Romo A, Sanchez-Tapia M, Lopez-Carrasco MG, Guillen-Pineda LE, Brito-Cordova GX, Martagon AJ, Granados-Portillo O, Walther G, Gomez-Perez FJ, Aguilar-Salinas CA, Tovar AR, Torres N, Almeda-Valdes P. Sucralose consumption modifies glucose homeostasis, gut microbiota, Curli protein, and related metabolites in healthy individuals: A randomized placebo-controlled, triple-blind trial. Clin Nutr ESPEN. 2025 Oct;69:733-744. doi: 10.1016/j.clnesp.2025.08.029. Epub 2025 Sep 2. PMID 40907790